CLINICAL TRIAL: NCT07318688
Title: A Randomized, Multicenter, Double-Blind, Placebo-Controlled Phase 3 Study to Evaluate the Efficacy and Safety of HMI-115 in Women With Moderate to Severe Endometriosis-Associated Pain Over a 24-Week Treatment Period and a 28-Week Extension
Brief Title: Evaluate the Efficacy and Safety of HMI-115 in Women With Moderate to Severe Endometriosis-associated Pain
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hope Medicine (Nanjing) Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HMI-115ENDO302
Record Dates: First submitted 2025-12-29; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Intervention Model Description: 1）Placebo-Controlled Double-blind Treatment Period (Week 0 to Week 24): Subjects will be randomized in a 1:1:1 ratio to receive subcutaneous (s.c.) injection with HMI-115 120 mg, HMI-115 240 mg or placebo every two weeks (Q2W). A total of 12 injections will be administered.
  2) Extension Treatment Period (Week 24 to Week 52): All eligible subjects who received placebo in the placebo-controlled double-blinded period will be randomized in a 1:1 ratio to receive HMI-115 120 mg Q2W or HMI-115 240 mg Q2W in the extension treatment period until Week 50, followed by an evaluation (Visit 29/EOT Visit) at Week 52. All eligible subjects in the active treatment groups will continue their treatment. A total of 14 injections will be administered.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- HMI-115_120mg (Experimental): 120mg, Once Every 2 weeks, subcutaneously injection,total of 26 injections (Week 0 to Week 52) or total of 14 injections (Week 24 to Week 52/Extension Treatment Period of Placebo )
  Interventions: Drug: HMI-115
- HMI-115_240mg (Experimental): 240mg, Once Every 2 weeks, subcutaneously injection,total of 26 injections (Week 0 to Week 52) or total of 14 injections (Week 24 to Week 52/Extension Treatment Period of Placebo )
  Interventions: Drug: HMI-115
- Placebo (Placebo Comparator): 2ml , Once Every 2 weeks, subcutaneously injection,total of 12 injections (Week 0 to Week 24)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HMI-115 — HMI-115 is human monoclonal antibody （120mg/vail）
  Arms: HMI-115_120mg; HMI-115_240mg
Drug: Placebo — Placebo （0mg/vail）
  Arms: Placebo

SUMMARY:
A phase 3 study to evaluate the efficacy and safety of HMI-115 in women with moderate to severe endometriosis-associated pain over a 24-week treatment period and a 28-week extension

ELIGIBILITY:
Inclusion Criteria:

* 1. Premenopausal female subjects, between 18 and 49 years of age, inclusive.
* 2. Has a surgical diagnosis of endometriosis (laparoscopy or laparotomy) as documented by medical records within 10 years before screening.
* 3. Has a Composite Pelvic Signs and Symptoms Score total score of ≥ 6 at screening with a score of at least 2 for DYS and at least 2 for NMPP.
* 4. Subject has reported "moderate" or "severe" for her endometriosis-associated DYS AND NMPP before randomization.
* 5. Subject has at least two consecutive regular menstrual cycle (i.e. 21 to 35 days in duration) prior to randomization.
* 6. Subject agrees to use required (nonhormonal) birth control methods during the entire length of participation in the study and agrees to avoid pregnancy from signing the informed consent until 12 weeks after the last dose.
* 7. Subject agrees to use only those rescue analgesic medications permitted by the protocol during the Screening, Treatment and Posttreatment follow-up Periods for her endometriosis-associated pain.
* 8. Criteria for Extension Treatment Period：Subject who completes treatment of the placebo-controlled double-blind treatment period and assessments at Week 24.

Exclusion Criteria:

* 1. Subject who is pregnant or breastfeeding or is planning a pregnancy during the study period or is less than 6 months post-partum or 3 months post-abortion at the time of entry into the Screening Period or pregnancy before randomization.
* 2. Subject has an intra-uterine device (IUD). Subject is eligible if she removes the IUD 1 month before screening.
* 3. Subject has chronic pelvic pain that is not caused by endometriosis (e.g., interstitial cystitis, irritable bowel syndrome) or has any other chronic pain syndrome (e.g., fibromyalgia, chronic back pain, myofascial pain syndrome, chronic headaches) that requires chronic analgesic or other chronic therapy, which would interfere with the assessment of endometriosis-associated pain.
* 4. Subject with a current history of undiagnosed abnormal genital bleeding.
* 5. Subject with history of hysterectomy and/or bilateral oophorectomy.
* 6. Subject has had surgery for endometriosis within 6 weeks prior to entry into the Screening Period.
* 7. Subject has previous history of a severe, life-threatening or other significant sensitivity to any opioids or non-steroidal anti-inflammatory drugs (NSAIDS) or any contraindication to their use such as gastrointestinal ulcer or bleeding.
* 8. Subject with known hypersensitivity to any of the IMP ingredients.
* 9. Subject has an estimated glomerular filtration rate (eGFR) of < 60mL/min/1.73 m2 at Screening Period.
* 10. Subject is currently participating in or has participated in an interventional clinical study with an investigational compound or device within 30 days prior to the start of Screening Period or 5 half-lives, whichever is longer.
* 11. Subject who has been exposed to HMI-115 treatment.
* 12. Subject has used medications such as hormones, analgesics, medications associated with bone loss, products that affect PRL levels, etc. within specific time window before Screening.
* 13. Subject has clinically significantly abnormal laboratory tests at Screening Period, including:

  1. Alanine transaminase (ALT/SGPT), or aspartate aminotransferase (AST/SGOT) ≥200% of the upper limit of normal, or total bilirubin (unless known diagnosis of Gilbert's syndrome) ≥ 150% of the upper limit of normal range.
  2. Hemoglobin < 100 g/L, Neutrophil count < 1.5×109/ L, Platelet count < 100×109/ L.
* 14. Subject has clinically significantly abnormal laboratory tests at Screening Period, including: Neutrophil count < 1.5×109/ L, Platelet count < 100×109/ L.
* 15. Subject has clinically significant abnormal ECG, or ECG with QTcF > 450 msec at Screening Period.
* 16. Subject has a history or current has malignancy except for treated basal cell carcinoma and cutaneous squamous cell carcinoma of the skin.
* 17. Subject is using any systemic corticosteroids for over 14 days within 3 months prior to Screening or is likely to require treatment with systemic corticosteroids during the study.
* 18. Subject has any of the following conditions within the last 6 months before Screening:

  1. Myocardial infarction, stroke, unstable angina or transient ischemic attack.
  2. Classified as being in New York Heart Association Class III or IV.
* 19. Subjects with body weight greater than 300 pounds or 136 kilograms.
* 20. Any other conditions in the Investigator's opinion that prevent the subject from participating.
* 21. Criteria for Extension Treatment Period： Subjects entering the follow-up period after treatment: subjects with a BMD decrease of ≥ 8.0% or Z-value ≤ -2.0 in any part of the lumbar spine, femoral neck, or total hip compared to baseline.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 540 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline (CFB) in dysmenorrhea (DYS) measured by Numeric Rating Scale (NRS) at Week 12 | week 12
CFB in non-menstrual pelvic pain (NMPP) measured by NRS at Week 12 | week 12

SECONDARY OUTCOMES:
CFB in DYS measured by NRS at Week 24 | week 24
CFB in NMPP measured by NRS at Week 12 | week 24
CFB in average overall pelvic pain measured by NRS at Week 12 and week 24 | Week 12 and week 24
CFB in DYSP measured by NRS at Week 12 and week 24 | Week 12 and week 24
Changes in the number of remedial analgesics allowed to be used compared to baseline | Week 12 and week 24
Adverse Events | During the clinical study period
  64 Weeks
To investigate the pharmacokinetics (PK) characteristic of HMI-115, Serum trough concentrations at each time point and descriptive statistics. | Before the first intervention、Week 2、Week 4、Week 8、Week 12、Week 16、Week 20、Week 24、Week 32、Week 40、Week 52
  Serum trough concentrations at each time point and descriptive statistics.
To investigate the immunogenicity of HMI-115：Anti-drug antibody (ADA) and Neutralizing antibody (NABs) | Before the first intervention、Week 2、Week 4、Week 8、Week 12、Week 16、Week 20、Week 24、Week 32、Week 40、Week 52

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Nanjing Women and children's healthcare hospital, Nanning, Jiangsu
  - Second Affiliated Hospital of Soochow University, Suzhu, Jiangsu
  - The International Peace Maternity and Child Health Hospital of the China Welfare Institute, Shanghai, Shanghai Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No